CLINICAL TRIAL: NCT05521802
Title: A Phase Ib/II Study of CBM.BCMA Chimeric Antigen Receptor T Cell Product (C-CAR088) for Treating Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of C-CAR088 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0203-029
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — B-Cell Maturation Antigen; bis(3-bis(4-chlorophenyl)methyl-4-dimethylaminophenyl)amine; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR088 (Experimental): Autologous C-CAR088 administered by intravenous (IV) infusion
  Interventions: Biological: B-cell maturation antigen (BCMA) directed chimeric antigen receptor (CAR)-T cell

INTERVENTIONS:
Biological: B-cell maturation antigen (BCMA) directed chimeric antigen receptor (CAR)-T cell — Autologous 2nd generation BCMA-directed CAR-T cells, single infusion intravenously

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and efficacy of C-CAR088 in patients with relapsed or refractory multiple myeloma. The phase Ib part of this study is to determine the recommended phase 2 dose (RP2D) of C-CAR088 in the targeted patient population.

DETAILED DESCRIPTION:
The study includes the following sequential procedures: Screening, Apheresis and C-CAR088 manufacturing, Baseline testing, Lymphodepletion, C-CAR088 infusion, and Follow-up Visit. Two dose levels of C-CAR088 will be tested during the phase Ib part to determine RP2D, which will be further evaluated during the phase II part.

ELIGIBILITY:
Inclusion Criteria

* ≥ 18 years of age, male or female patients
* Relapsed or refractory multiple myeloma
* Have been treated with ≥ 3 prior lines of therapy, including at least one proteasome inhibitor and one immunomodulatory drug, and had progressed during or within 12 months post the last treatment.
* Had measurable disease as defined by any of the following criteria:

  * Serum M protein ≥ 0.5g/dL
  * Urine M protein ≥ 200mg/24h
  * Serum free light chain (sFLC): abnormal κ/λ ratio with involved sFLC ≥ 100mg/L
* Adequate liver, renal, bone marrow, and heart function
* Eastern cooperative oncology group (ECOG) 0-1

Exclusion Criteria

* Any known allergies to the components or excipients of the C-CAR088 cell product
* Prior allogeneic hematopoietic stem cell transplantation (HSCT) at anytime, or autologous stem-cell transplantation (ASCT) within 12 weeks prior to apheresis
* Central nervous system (CNS) involvement
* Stroke or convulsion history within 6 months prior to signing informed consent form (ICF)
* Plasma leukemia
* Autoimmune disease, immunodeficiency or diseases requiring immunosuppressants treatment
* Uncontrolled active infection; active hepatitis B virus (HBV), hepatitis C virus (HCV) infection; HIV or syphilis infection
* Severe heart, liver, renal or metabolism disease
* Inadequate wash-out time for previous anti-tumor treatments prior to apheresis
* Previous CAR-T cell treatment, genetically modified T-cell therapies or BCMA-directed treatment history
* History or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's safe participation and compliance in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
[phase Ib] Incidence and severity of Adverse Events | 24 months
  Incidence and severity of Adverse Events
[phase II] Overall response rate (ORR) at 3 months after C-CAR088 infusion | 3 months
  the rate of patients with best response of partial response (PR) or better at 3 months after C-CAR088 infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | 24 months
  The rate of patients with best response of partial response (PR) or better
[phase Ib] Overall response rate (ORR) at 3 months after C-CAR088 infusion | 3 months
  The rate of patients with best response of partial response (PR) or better at 3 months after C-CAR088 infusion
Duration of response (DOR) | 24 months
  The time from the first documented PR or better response to relapse or death, whichever occurs first
Time to response (TTR) | 24 months
  The time from the date of C-CAR088 infusion to the first documented PR or better
Progression-free survival (PFS) | 24 months
  The time from the date of C-CAR088 infusion to the date of first documented disease progression or death
Overall survival (OS) | 24 months
  The time from the date of C-CAR088 infusion to the date of death
Minimal residual disease (MRD) negativity rate | 24 months
  The rate of patients reached MRD negativity
[phase II] Incidence and severity of Adverse Events | 24 months
  Incidence and severity of Adverse Events
Maximal plasma concentration (Cmax) | 24 months
  maximal plasma concentration of C-CAR088 in peripheral blood
Time to reach the maximal plasma concentration (Tmax) | 24 months
  Time to reach the maximal plasma concentration of C-CAR088 in peripheral blood
Area under the curve within 28 days (AUC0-28d) | 28 days
  Area under the curve of C-CAR088 in peripheral blood within 28 days post infusion
Time of last measurable observed concentration (Tlast) | 24 months
  Time of last measurable observed concentration of C-CAR088 in peripheral blood
Anti-drug (C-CAR088) antibody | 24 months
  Presence of serum anti-drug (C-CAR088) antibody
Serum M protein | 24 months
  serum M proteins concentration changes over time
Urine M protein | 24 months
  Urine M proteins concentration changes over time
Serum free light chain (sFLC) | 24 months
  Serum free light chain (sFLC) concentration changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Tianjin, China